CLINICAL TRIAL: NCT00558558
Title: A Phase II Study Examining the Role of Fermented Soy Beverage for Improving Cancer-Associated Anorexia and Cachexia
Brief Title: Haelan and Nutrition in Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to low recruitment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Haelan Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0370
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Results first posted 2011-10-12 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2011-09

CONDITIONS: Anorexia; Weight Loss; Cachexia
Keywords: Solid Tumors; Cancer-Associated Anorexia; Weight Loss; Haelan; Fermented Soy Product; Nutrition; Cachexia
MeSH Terms: conditions — Anorexia; Weight Loss; Cachexia | interventions — Flurandrenolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fermented Soy Supplement (Other): 4 oz Haelan orally twice daily for 8 weeks
  Interventions: Drug: Haelan

INTERVENTIONS:
Drug: Haelan — 4 oz orally twice daily for 8 Weeks
  Other Names: Fermented Soy Supplement

SUMMARY:
Primary:

* To determine if treatment with Haelan (fermented soy product) can decrease the severity of poor appetite measured using a visual analog scale (VAS) of 0 to 100 mm (0 mm = best, 100 mm = worst) at week 4 +/- 5 days.
* To determine if treatment with Haelan can decrease the severity of nausea, fatigue, and improve patients' overall sense of well being measured using a VAS of 0 to 100 mm (0 mm = best, 100 mm = worst) at week 4 +/- 5 days.
* To determine if treatment with Haelan can increase patient's calorie intake, albumin, pre-albumin, anthropometric measure, lean body mass (measured by bio-impedence analysis), and weight at week 4+/- 5 days.
* To determine if treatment with Haelan can decrease patient's Functional assessment of anorexia/cachexia therapy subscales or (FAACT) and the Functional Assessment of Chronic Illness Therapy with fatigue subscales (FACIT-F) at week 4+/- 5 days.
* To assess the feasibility of accrual, and adherence to the Haelan consumption.

Secondary:

* Determine the plasma isoflavone activity, 12-MTA and 13-MTA of these patients.
* Correlate the biologic modulation of peripheral blood lymphocyte NF-kB by Haelan with primary outcome in these patients.
* To determine if treatment with Haelan can increase patient's functional status at week 4+/- 5 days.

DETAILED DESCRIPTION:
Individuals who have cancer-related malnutrition have also been found to have a higher risk of complications and are less able to tolerate the side effects of conventional therapies such as chemotherapy, radiation, and surgery.

Haelan is a soy-based liquid (beverage). It contains large amount of isoflavones. Isoflavones inhibit "nuclear factor-kappa B," which may lead to prevention of weight loss.

If you are eligible to take part in this study, you will then be given 2 fluid ounces of Haelan, as a taste test. If you are not able to tolerate the taste of Haelan, you will not be eligible for this study.

If you are able to pass the taste test and you are a woman who is able to have children, you will be asked to have a pregnancy test 24 hours prior to registration to Part B. Then only if you test negative for the pregnancy test will you be considered eligible for this study. If you are a female patient and refuse to practice accepted methods of contraceptives during the study, you will not be eligible for this study.

If you are still eligible for this study, you will have about 6 teaspoons of blood drawn, for baseline routine tests. Your height and weight will be measured. You will be instructed by a research nurse to recall your one day food intake before starting treatment. You will be asked about any medications you are taking (especially any appetite stimulants, such as megestrol, corticosteroid, and marinol), including the dose and when you take them. If you are able to tolerate the taste of Haelan, you will be instructed to drink 4 ounces of Haelan soy beverage 2 times a day, on an empty stomach, for 8 weeks. You may add water, stevia, honey or artificial sweeteners into Haelan prior to drinking it to improve the tolerance of Haelan. If you are unable to tolerate 4 ounces of Haelan twice a day after 2 attempts, the dose will be reduced to 2 ounces twice a day. If you are still not able to tolerate it after 2 attempts, the dose will be reduced again to 1 ounce twice a day. If you still cannot tolerate drinking this Haelan dose after 2 more attempts, the dose will be reduced again to 1 ounce daily. If you cannot tolerate at least 1 ounce a day for 5 consecutive days, you will be taken off this study. If you vomit within half hour of taking the Haelan, you should try at least 2 more times to drink at least 1 ounce of Haelan on the same day. If unsuccessful, please record that you were not able to take the Haelan on that day. If you cannot tolerate at least 1 ounce of Haelan a day for 5 days in a row, you will be taken off this study.

If you are able to pass the taste test and if you are a female with child-bearing potential you will be asked to have a pregnancy test 24 hours prior to registration to Part B .

You will be asked to write down how many ounces of Haelan you are able to drink at each dose and each day, in a study-drug diary. You will be asked to write down the side effect of Haelan daily.

You will be asked to write down the side effect of Haelan daily. You will have about 6 teaspoons of blood drawn for routine clinical tests, for protein level and kidney function at Week 4 +/- 5 days. You will also be asked to complete 3 questionnaires that have questions about any appetite, nausea, and fatigue you experience and your overall sense of well being. These questionnaires will take about 15 minutes to complete. You will be given several tests to measure your weight, skin-fold thickness and body composition. You will be given 2 functional tests, which involves timing how long it takes for you to get up from a chair to walk and timing how long it takes for you to walk 50 feet at your fastest speed. These tests will take about 30 minutes to complete. The questionnaires, measurement of your weight, skin-fold thickness and body composition, and functional tests will be done before treatment starts and on a visit day 10 +/- 5 days, week 4 +/- 5 days, week 6 +/- 5 days.

You will also be instructed by a research nurse to record your food intake, for one day in day 10 +/- 5 days, week 4 +/- 5 days, week 6 +/- 5 days.

During this study, you will have several tests performed to check for safety and effectiveness. Every 2 weeks, you will be asked if you are experiencing any side effects, either related or not related to the treatment. You will be asked about any medications you are taking, including the dose levels and when you take them.

You will be asked to bring the Haelan intake diary back to clinic on the study visits between day 10 +/- 5 days, week 4 +/- 5 days, week 6 +/- 5 days, so the study staff can record how many ounces of Haelan you have taken every day.

At the end of Haelan soy beverage treatment (week 8 +/- 5 days), you will be asked to return to the clinic for a end-of-treatment visit. You will have blood drawn (about 6 teaspoons) for routine clinic tests to detect for protein level and kidney function. Your study-drug diary will be checked, and you will again be given the questionnaires. Measurement of your weight, skin-fold thickness and body composition, and functional tests will be given. You will be asked about any medications you are taking, including the dose levels and when you take them. You will also be asked to provide the research nurse with the record of one day food intake at 8 weeks +/- 5 days. The one day food intake record should be finished before coming in for your clinic visit, as long as it is the recording of the 8th week food intake. However, if the 8th-week clinic visit is on the first day of the 8th week, you can continue to record your food intake after the visit, and then return it to the research nurse at a later time. For this record, you need to write down what type of food you eat, and the estimated portion (for example: rice, 2 ounces; slice of apple pie, 1/8 of a pie).

If you are currently taking megestrol, any corticosteroid, mirtazapine, metoclopramide, or dronabinol and you change your dose while on study, you will be taken off study. Also, if you were not on them before but you start taking any of the above listed drugs while on this study, you will be taken off study.

This is an investigational study. About 32 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Anorexia (defined as > 30mm on a visual analog scale [VAS] of 0 to 100mm)
2. Weight loss (defined as weight loss > 5% within last 6 months)
3. Normal cognition (per treating physician's opinion)
4. Written informed consent
5. Advanced solid tumor (defined as locally recurrent or metastatic disease)
6. Patient must have perceived weight loss as a problem.
7. Able to maintain oral food intake within one week prior to enrollment in this study.

Exclusion Criteria:

1. Evidence of ascites (per treating physician's opinion).
2. Receiving supplementary tube feedings or parenteral nutrition
3. Known mechanical obstruction of the alimentary tract, or intractable vomiting
4. Add or change dose of the following medication within 2 weeks prior to this trial or during this trial: megestrol, corticosteroid, mirtazapine, metoclopramide and dronabinol, with the exception of pre-medication for chemotherapy (10-20 mg Decadron intavenous (IV) once and/or Reglan 10 mg IV x1 prior to chemotherapy).
5. Allergic to soy.
6. Positive pregnancy test for female patients of child-bearing potential. (Definition of child-bearing potential: not post-menopausal for past 12 months or nor surgically sterile)
7. Female patients with child bearing potential, but refuse to practice accepted methods of contraception (acceptable forms of contraception include: continuous abstinence, Depo-Provera shot, tubal ligation, NuvaRing vaginal ring, Ortho Evra skin patch, oral contraceptive, IUD-Mirena, vasectomy, male condom, diaphragm).
8. Weight less than 80 lb.
9. Patient who could not tolerate oral intake of 2 Oz. of Haelan during the taste test.
10. Diagnosed of breast cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 10/22/07 to 07/24/08. All patients recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the six patients registered, two patients were ineligible and not included in any group assignment. Four patients were not eligible for analysis.
Period: Overall Study
Arm/Group | Fermented Soy Supplement
Started | 6
Completed | 0
Not Completed | 6
Not completed — Unable to swallow | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Fermented Soy Supplement
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 59 [50 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Poor Appetite Following Treatment With Haelan (Fermented Soy Product)
Description: Change in severity of poor appetite measured using a visual analog scale (VAS) of 0 to 100 mm (0 mm = best, 100 mm = worst) at week 4 +/- 5 days.
Time Frame: Baseline and Week 4 +/- 5 days
Population: The participants were not eligible for analysis based on the primary outcome timeline.
Arm/Group | Fermented Soy Supplement
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Fermented Soy Supplement
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fermented Soy Supplement (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No